CLINICAL TRIAL: NCT04443088
Title: A Phase 1a/1b, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Evidence of Antitumor Activity of INV-1120 As a Single Agent and in Combination with Pembrolizumab in Adult Patients with Advanced Solid Tumors
Brief Title: An Open-Label Study of INV-1120 As a Single Agent and in Combination with Pembrolizumab in Adult Patients with Advanced Solid Tumors
Acronym: KEYNOTE-E12
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Ionova Life Sciences Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INV-1120-101(MK-3475-E12)
Record Dates: First submitted 2020-05-29; First posted 2020-06-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Solid Tumor, Adult; Cancer Metastatic; Solid Carcinoma; Solid Tumor, Unspecified, Adult; Tumor, Solid
Keywords: Ionova; Ionova Bio; Cancer; Oncology
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation (Other): Phase 1a: Subjects will receive escalating doses of INV-1120 orally once a day until un-acceptable toxicity or disease progression. Three to six patients will be enrolled per cohort to evaluate the safety and pharmacokinetics for each dose level. After the last patient in each cohort completes Cycle 1 (DLT observation period of 28 days), the Safety Evaluation Team (SET) will evaluate the safety data and pharmacokinetic collected from Cycle 1, and make the decision whether to escalate the dose before opening the second cohort.
  Phase 1b: Subjects will receive escalating and de-escalating doses of INV-1120 orally once a day in combination with pembrolizumab until un-acceptable toxicity or disease progression, and DLT observation period of 21 days.
  Interventions: Drug: INV-1120; Combination Product: Pembrolizumab

INTERVENTIONS:
Drug: INV-1120 — INV-1120 is an investigational selective and potent small molecule indicated for the treatment of solid malignancies including, but not limited to colorectal, breast, pancreatic, lung and liver cancers.
Combination Product: Pembrolizumab — Pembrolizumab will be administered as a dose of 200 mg on Day 1 of each 3-week treatment cycle.
  Other Names: KEYTRUDA®

SUMMARY:
Phase 1, open-label dose-escalation study to determine the MTD of INV-1120 and RP2D, and to assess the DLT of INV-1120 as a single agent or in the combination with pembrolizumab. The safety, tolerability, and PK of INV-1120 as a single agent or in the combination with pembrolizumab will be assessed in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
Phase 1a: it is anticipated that approximately 36 patients will be enrolled in the dose escalation phase as a single agent of the study. Additionally, up to 9 additional patients may be enrolled to confirm the safety of patients treated at the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D).

Phase 1b: approximately 36-42 patients will be enrolled in the dose escalation and de-escalation phases in the combination with pembrolizumab. One or more combination dose levels that could represent the combination RP2D will be expanded to a total of 12-15 patients to confirm safety and tolerability of the combination.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, according to local guidelines, signed and dated by the patient prior to the performance of any study-specific procedures, sampling, or analyses;
2. Patient must be ≥18 years-of-age at the time of signature of the informed consent form (ICF);
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1;
4. Patients with histologically or cytologically confirmed advanced solid tumors which have progressed on or following standard therapy or for which no standard therapy exists;
5. Patients with life expectancy ≥3 months;
6. Patients with at least one measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI), according to RECIST v1.1. Tumor lesions that have been irradiated ≥4 weeks before the start of treatment, and have subsequently had documented progression, may be chosen as target lesions in the absence of measurable lesions that have not been irradiated;
7. Patients whose laboratory data at screening meet the acceptable criteria for bone marrow, liver function and renal function.
8. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test during screening. A woman is considered of childbearing potential (fertile) following menarche and until becoming postmenopausal unless permanently sterile. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. Postmenopausal women can be included;
9. Male patients with female partners of childbearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 3 months following last dose. Medically acceptable contraception includes:

   * Hormonal methods (Needs to have been instituted at least 1 month prior to the first dose of study drug):
   * Barrier methods:
   * Abstinence, defined as refraining from sexual intercourse
10. Male patients must also refrain from donating sperm from the first dose of study drug until 4 months after the last dose of study drug;
11. Patients must be able to swallow and retain orally administered medication.

Exclusion Criteria:

1. History (≤5 years) or current evidence of cancer that is histologically distinct from the cancer under study, except for cervical carcinoma in situ, superficial non-invasive bladder tumors, or curatively treated Stage I non-melanoma skin cancer. Patients with hepatocellular carcinoma will be excluded from Phase 1b dose escalation;
2. Known serious allergy to investigational drug or excipients (microcrystalline cellulose);
3. History of severe autoimmune disease (including significant ongoing immune-related adverse events of prior immune-oncology therapy) or autoimmune disorder that requires chronic systemic corticosteroid treatment at immunosuppressive doses (prednisone >10 mg/day or equivalent);
4. Known malignant central nervous system disease other than neurologically stable, treated brain metastases - defined as metastases having been treated by surgery, surgery plus radiotherapy or radiotherapy alone, with no evidence of progression or hemorrhage and off any systemic corticosteroids for at least 4 weeks prior to signing the consent;
5. History (within 4 weeks of starting treatment) or evidence of active infections (Grade ≥2);
6. Seropositive status for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at any time before the start of treatment: Testing for seropositive status during screening will be at the discretion of the Investigator in patients without previously reported results;
7. History or evidence of any severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the Investigator and Sponsor, could affect the patient's participation in the study, such as any disorder or surgical procedure that could impact the absorption of study drug from the gastrointestinal tract.
8. History (≤6 months before the start of treatment) or evidence of any of the following: acute myocardial infarction, unstable angina pectoris, coronary artery bypass graft, cerebrovascular accident, or transient ischemic attack;
9. Patients who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * Congenital long QT syndrome;
   * Significant ventricular or supraventricular arrhythmias (patients with sinus arrhythmia or chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible);
   * LVEF < 50% by ECHO or MUGA;
   * Other clinically significant heart disease such as known congestive heart failure New York Heart Association (NYHA) Class III-IV;
10. Patients with QT interval ≥470 msec in females and ≥450 msec in males at screening using Fridericia's formula (determined as the mean of 3 QTcF values from the screening triplicate ECG obtained with adequate quality);
11. Women who are pregnant or breastfeeding.
12. WOCBP and sexually active fertile men with WOCBP partners who are unwilling or unable to use acceptable contraception method to avoid pregnancy for at least 1 month before the first dose of the study drug, during the study, and for 4 months after the last dose of study drug;
13. Male patient who plans to father a child while enrolled in this study or within 4 months after the last dose of study drug;
14. Not recovered from toxicity from prior anticancer therapy to baseline or Grade 1 (except toxicities which are not clinically significant such as alopecia, skin discoloration).
15. History of an allogeneic bone marrow or solid organ transplant;
16. Use of systemic anti-cancer agent (except luteinizing hormone-releasing hormone (LHRH) agonists, bisphosphonates and denosumab) or investigational drug ≤28 days or five half-lives whichever is shorter prior to the first dose of study treatment;
17. Radiation therapy ≤28 days prior to the first dose of study treatment, or likely to require radiation therapy at any time until the 30 days after the last dose of study treatment, except for palliative radiation therapy limited to non-target bone lesions;
18. Major surgery within 4 weeks before enrollment or surgery with ongoing post-operative complications);
19. History of transfusion of platelets ≤2 weeks before the start of treatment;
20. Patients who start erythropoietin or granulocyte-colony stimulating factor (G-CSF), pegfilgrastim, or filgrastim ≤3 weeks before screening;
21. Patients taking medications known to have a significant risk of causing Torsades de Pointes. Patients who have discontinued any of these medications must have a wash-out period of at least 7 days or at least 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug.
22. History of use of H2 blockers (<24 hours before the first dose of study treatment and during the study) and proton pump inhibitors (<5 days before the first dose of study treatment and during the study).
23. Patients with recent (within past 12 months) history, or are currently being treated for gastroesophageal ulcer.

    The following additional exclusion criteria will apply to patients enrolling in Phase 1b:
24. Have been discontinued treatment due to a Grade 3 or higher immune-related (irAE) from prior anti-PD-1 or anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137) (only for dose expansion).
25. Patient is currently participating or has participated in a study of an investigational agent or using an investigational device within 30 days of administration of investigational products.
26. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Note: Administration of killed vaccines are allowed.
27. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
28. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease or radiation pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Determine DLTs and RP2Ds in INV-1120 | 12 months
  To evaluate dose limiting toxicities (DLTs) of INV-1120 in patients with advanced cancer and to establish a recommended Phase 2 dose (RP2D)
Phase 1b: Determine RP2D and DLTs of the combination of INV-1120 and pembrolizumab | 12 months
  To determine RP2D, and to assess DLT of the combination of INV-1120 and pembrolizumab administered to adult patients with advanced solid tumors.

SECONDARY OUTCOMES:
Phase 1a: Determine the PK using AUC of INV-1120 | 12 months
  To determine the pharmacokinetics (PK) using AUC of INV-1120 after a single dose and at steady state after multiple doses
Phase 1b: Determine the PK using AUC of INV-1120 | 12 months
  To determine the pharmacokinetics (PK) using AUC of INV-1120 after a single dose and at steady state after multiple doses in combination with pembrolizumab
Phase 1a: Determine the PK using Cmax of INV-1120 | 12 months
  To determine the pharmacokinetics (PK) using Cmax of INV-1120 after a single dose and at steady state after multiple doses
Phase 1b: Determine the PK using Cmax of INV-1120 | 12 months
  To determine the pharmacokinetics (PK) using Cmax of INV-1120 after a single dose and at steady state after multiple doses in combination with pembrolizumab
Characterize investigator defined response overall response rate (ORR) etc using RECIST v1.1 | 12 months
  To characterize Investigator defined ORR, PFS and DOR using RECIST v1.1
Phase 1a: Characterize the safety of INV-1120 as assessed by CTCAE v5.0 | 12 months
  To analyze the safety profile of INV-1120 as a single agent by AE, clinical lab test results, ECG and Vital signs changes
Phase 1b: Characterize the safety of the combination of INV-1120 and pembrolizumab as assessed by CTCAE v5.0 | 12 months
  To analyze the safety profile of the combination of INV-1120 and pembrolizumab by AE, clinical lab test results, ECG and Vital signs changes

OTHER OUTCOMES:
Phase 1a: Characterize investigator defined ORR using iRECIST | 12 months
  To characterize investigator defined ORR using iRECIST
Phase 1a: Characterize investigator defined PFS using iRECIST | 12 months
  To characterize investigator defined PFS using iRECIST
Phase 1a: Characterize investigator defined DOR using iRECIST | 12 months
  To characterize investigator defined DOR using iRECIST

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Horizon Oncology Research, LLC,, Lafayette, Indiana
  - START, San Antonio, Texas
  - UT Health, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No